CLINICAL TRIAL: NCT00177528
Title: Safety and Efficacy of Venlafaxine XR in Elderly Patients With Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000918
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-10

CONDITIONS: Depression
Keywords: Elderly
MeSH Terms: conditions — Depression

INTERVENTIONS:
Drug: venlafaxine-XR

SUMMARY:
This research study is to evaluate the safety and usefulness of venlafaxine-XR in the treatment of major depression in the elderly.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to evaluate the safety of venlafaxine extended release formulation (XR) in the treatment of geriatric non-psychotic depression. This pilot study's specific aims are to assess the safety of venlafaxine XR in the geriatric population, to estimate the response rate of older depressed subjects treated under open conditions and to evaluate pharmacokinetic characteristics that may impact on safety and outcome.

ELIGIBILITY:
Inclusion Criteria:

* men and women of all races who are 60 years old or older;
* a DSM-IV diagnosis of major depressive episode without psychotic features;
* 17-item Ham-D score of >15 for potential subjects who have not received any antidepressant treatment during this illness episode or HAM-D > 11 for potential subjects who have received treatment with an antidepressant (other than venlafaxine-XR) during this illness episode;
* a MMSE score of >15.

Exclusion Criteria:

* history of meeting DSM-IV criteria for mania, schizophrenia or other psychotic disorder;
* history of substance abuse or dependence, including alcohol, within the last three months;
* current hyponatremia (as defined as a serum sodium level < 130 meq/l);
* untreated or uncontrolled hypertension;
* a history of being unable to tolerate venlafaxine-XR or venlafaxine immediate release formulation;
* history of receiving venlafaxine-XR or venlafaxine immediate release formulation of 6 or more weeks at 300mg/d during index depressive episode; (7) EKG revealing QTc > 480 msec;
* myocardial infarction, unstable angina, palpitation or cardiogenic syncope within 3 months prior to entering this study;
* the presence of active suicidal ideation with intent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2000-10; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of venlafaxine XR.
Rate of Major Depression remission to treatment.

SECONDARY OUTCOMES:
Participant characteristics that influence safety and remission rate.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Whyte, MD, Principal Investigator — University of Pittsburgh; Benoit H Mulsant, MD, Principal Investigator — University of Pittsburgh; Charles F. Reynolds III, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States